CLINICAL TRIAL: NCT06685913
Title: The Effect of Ketone Esters on Forearm Glucose Metabolism
Acronym: KAV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 5390017
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Blood glucose; Ketone monoester; Substrate metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Coded, known only to one independent individual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone supplementation (Experimental): 100 mL flavoured drink containing 0.3 g/kg ketone monoester ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate; ΔG®, University of Oxford; https://www.deltagketones.com)
  Interventions: Dietary Supplement: Ketone supplement
- Placebo (Placebo Comparator): Placebo with bitter agent to flavour match
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Ketone supplement — 100 mL flavoured drink containing 0.3 g/kg ketone monoester ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate; ΔG®, University of Oxford; https://www.deltagketones.com) consumed 30 min prior to a mixed meal tolerance test
  Arms: Ketone supplementation
Dietary Supplement: Placebo supplement — Placebo with bitter agent to flavour match, consumed 30 min prior to a mixed meal tolerance test
  Arms: Placebo

SUMMARY:
Ketones are naturally produced by our body and can affect our blood sugar levels. Ketones could be important tool for treating disease or recovering from exercise. The purpose of this research is to determine if a ketone drink can increase sugar uptake in our muscles. This research will provide new knowledge about the regulation of blood sugar.

DETAILED DESCRIPTION:
Impaired skeletal muscle glucose uptake following a meal ("insulin resistance"), is a primary risk factor for developing type 2 diabetes. We and others have consistently shown that ingesting exogenous ketones can reduce blood glucose concentration. Mechanistically, this must arise through reduced glucose release (i.e. from liver), and/or increased uptake (i.e. into skeletal muscle). Our current MRC-funded work is focussing on ketone-liver interactions in patients with type 2 diabetes. Here we aim to investigate how KE influence skeletal muscle glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40

Exclusion Criteria:

* Any diagnosed metabolic health condition
* Pregnant
* Smoker
* Diagnosed Cardiovascular disease
* Use of medications deemed by research team to affect study outcomes
* Recent history of musculoskeletal injury
* Aged >40 or <18
* Allergy to ingredients in the supplement, including ketones, lactose or milk protein

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Forearm glucose net balance | 3 hours
  Net balance of blood glucose across a forearm following a mixed meal tolerance test

SECONDARY OUTCOMES:
Forearm non-esterified fatty acid net balance | 3 hours
  Net balance of blood non-esterified fatty acids across a forearm after a mixed meal tolerance test
Forearm amino acid net balance | 3 hours
  Net balance of blood amino acids across a forearm following a mixed meal tolerance test
Serum insulin concentrations | 3 hours
  Insulin concentration using ELISA assay over 4 and 8 hours following a meal
Ketone concentration | 3 hours
  Ketone concentration using colorimetric assay over 4 and 8 hours following a meal

CONTACTS AND LOCATIONS:
Overall Officials: George F Pavis, PhD, Principal Investigator — University of Exeter
Locations (1):
- Nutritional Physiology Research Unit, University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on open access public repositories
Supporting Information: Study Protocol, SAP, CSR